CLINICAL TRIAL: NCT06986512
Title: Rapid Detection of Pseudomonas Aeruginosa in Bronchoalveolar Lavage Fluid Using Label-free Single-particle Imaging Technology and Assessment of Post-treatment Efficacy in Patients With Pseudomonas Aeruginosa Infection
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-806
Record Dates: First submitted 2025-03-11; First posted 2025-05-23 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-05

CONDITIONS: Rapid Detection; Pseudomonas Aeruginosa Infection
MeSH Terms: conditions — Pseudomonas Infections | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — The investigators will dynamically and continuously collect bronchoalveolar lavage fluid samples from participants and diagnosed with Pseudomonas aeruginosa infection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bronchoscopy — We will perform bronchoscopy and collect bronchoalveolar lavage fluid (BALF)

SUMMARY:
The aim of this study is to observe specimens of bronchoalveolar lavage fluid from patients using a reflection enhanced dark-field scattering microscopy. By observing parameters such as the size, morphology, scattering intensity, and movement speed of pathogens, combined with the clinical characteristics of patients, a rapid diagnosis of Pseudomonas aeruginosa infection can be made. At the same time, the bronchoalveolar lavage fluid samples of patients infected with Pseudomonas aeruginosa before and after treatment were compared, and the quantity and vitality of Pseudomonas aeruginosa were observed to judge the efficacy of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* After admission, Pseudomonas aeruginosa was cultured in bronchoalveolar lavage fluid or lower respiratory tract aspirates

Exclusion Criteria:

* Age under 18 years old or over 90 years old
* Pregnancy, lactation period -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected or diagnosed patients with pulmonary infection caused by Pseudomonas aeruginosa
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The size of pathogens | From enrollment to the end of treatment at 2 weeks
  Measure the size of pathogens
scattering intensity of pathogen | From enrollment to the end of treatment at 2 weeks
  Determine the shape of pathogens through scattering intensity
movement speed of pathogens | From enrollment to the end of treatment at 2 weeks
  Measure the movement speed of pathogens, such as flagellates like Pseudomonas aeruginosa, which have a fast movement speed

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China